CLINICAL TRIAL: NCT01389765
Title: Effect of Food on the Pharmacokinetics of LY2216684 in Healthy Subjects
Brief Title: A Study to Evaluate the Effect of Food on LY2216684
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 12620; H9P-EW-LNDC (Other: Eli Lilly and Company)
Record Dates: First submitted 2011-07-06; First posted 2011-07-08 (Estimated); Results first posted 2018-11-13 (Actual); Last update posted 2018-11-13 (Actual); Status verified 2018-11

CONDITIONS: Depressive Disorder, Major
MeSH Terms: conditions — Depressive Disorder, Major | interventions — alpha-((5-fluoro-2-methoxyphenyl)methyl)-alpha-(tetrahydro-2H-pyran-4-yl)-2-morpholinemethanol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- LY2216684 administered in fasted then fed state (Experimental): Period 1: Single 18-mg (milligram) oral dose of LY2216684 administered in fasted state. Period 2: Single 18-mg oral dose of LY2216684 administered in fed state. Periods will be separated by a minimum of 7 days.
  Interventions: Drug: LY2216684
- LY2216684 administered in fed then fasted state (Experimental): Period 1: Single 18-mg oral dose of LY2216684 administered in fed state. Period 2: Single 18-mg oral dose of LY2216684 administered in fasted state. Periods will be separated by a minimum of 7 days.
  Interventions: Drug: LY2216684

INTERVENTIONS:
Drug: LY2216684 — Administered orally

SUMMARY:
This study will evaluate the effect of food on LY2216684. There will be 2 study periods each lasting up to 5 days. There will be at least 7 days between the two doses and a follow up will occur at least 7 days after the last dose. Screening is required within 30 days prior to the start of the study.

ELIGIBILITY:
Inclusion Criteria:

* Male subjects: Agree to use a reliable method of birth control during the study and for 1 month following the last dose of study drug.
* Female subjects: Are women of child-bearing potential who test negative for pregnancy at the time of enrollment, have used a reliable method of birth control for 4 weeks prior to administration of study drug, and agree to use a reliable method of birth control during the study and for 1 month following the last dose of study drug; or women not of child-bearing potential due to surgical sterilization (hysterectomy, bilateral oophorectomy, or tubal ligation) or menopause [at least 1 year without menses or 6 months without menses and a follicle stimulating hormone (FSH) >40 mIU/mL (milli-international-units/milliliter)]
* All Subjects:

  * Are overtly healthy as determined by medical history and physical examination
  * Have a body weight >50 kg (kilogram)
  * Have clinical laboratory test results within normal reference range for the population or investigator site, or results with acceptable deviations that are judged to be not clinically significant by the investigator
  * Have venous access sufficient to allow for blood sampling as per the protocol
  * Are reliable and willing to make themselves available for the duration of the study and are willing to follow study procedures
  * Have given written informed consent approved by Lilly and the institutional review board (IRB) governing the site
  * Have normal blood pressure (BP) and pulse rate (sitting position)
  * Are willing to eat all components in the standard high-fat meal

Exclusion Criteria:

* Are currently enrolled in, have completed or discontinued within the last 30 days from, a clinical trial involving an investigational product other than the investigational product used in this study; or are concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study
* Have known allergies to LY2216684, related compounds, or any components of the formulation
* Are persons who have previously received the investigational product in this study, have completed or withdrawn from this study or any other study investigating LY2216684 within 6 months prior to Screening
* Have an abnormality in the 12-lead electrocardiogram (ECG) that, in the opinion of the investigator, increases the risks associated with participating in the study
* Have a history of suicidal ideation or suicide attempts
* Have a history of/or current cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; of constituting a risk when taking the study medication; or of interfering with the interpretation of data
* Regularly use known drugs of abuse and/or show positive findings on urinary drug screening
* Show evidence of human immunodeficiency virus (HIV) infection and/or positive human HIV antibodies
* Show evidence of hepatitis C and/or positive hepatitis C antibody
* Show evidence of hepatitis B and/or positive hepatitis B surface antigen
* Are women with a positive pregnancy test or women who are lactating
* Intend to use over-the-counter or prescription medication within 14 days prior to dosing unless deemed acceptable by the investigator and sponsor's medical monitor, except for influenza vaccinations
* Have donated blood of more than 500 mL (milliliter) within the last month
* Have an average weekly alcohol intake that exceeds 21 units per week (males) or 14 units per week (females), or are unwilling to stop alcohol consumption from 48 hours prior to dosing in each period until discharge in each period [1 unit = 12 oz (ounces) or 360 mL of beer; 5 oz or 150 mL of wine; 1.5 oz or 45 mL of distilled spirits]
* Consume 5 or more cups of coffee (or other beverages or foods of comparable caffeine content) per day, on a habitual basis, or are unwilling to stop caffeine consumption from 48 hours prior to dosing in each period until discharge in each period
* Subjects must adhere to the smoking restrictions of the Clinical Research Unit (CRU) while a resident of the CRU
* Have consumed grapefruit or grapefruit-containing products, starfruit, or pomegranates 7 days prior to enrollment or are unwilling to avoid them during the study
* Subjects determined to be unsuitable by the investigator for any reason
* Have a documented or suspected history of glaucoma

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2011-07; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Daytona Beach, Florida, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- LY2216684 During Fed, Then LY2216684 During Fasting State: In Period 1, participants received a single oral dose of 18 milligram (mg) LY2216684, administered in fed state. In Period 2, participants received a single oral dose of 18 mg LY2216684, administered in the fasting state. Periods were separated by a 7-day washout period.
- LY2216684 During Fasting, Then LY2216684 During Fed State: In Period 1, participants received a single oral dose of 18 milligram (mg) LY2216684, administered in fasting state. In Period 2, participants received a single oral dose of 18 mg LY2216684, administered in the fed state. Periods were separated by a 7-day washout period.
Period: First Intervention (Day 1)
Arm/Group | LY2216684 During Fed, Then LY2216684 During Fasting State | LY2216684 During Fasting, Then LY2216684 During Fed State
Started | 12 | 12
Completed | 12 | 12
Not Completed | 0 | 0
Period: Washout Period (7 Days)
Arm/Group | LY2216684 During Fed, Then LY2216684 During Fasting State | LY2216684 During Fasting, Then LY2216684 During Fed State
Started | 12 | 12
Completed | 12 | 12
Not Completed | 0 | 0
Period: Second Intervention (Day 1)
Arm/Group | LY2216684 During Fed, Then LY2216684 During Fasting State | LY2216684 During Fasting, Then LY2216684 During Fed State
Started | 12 | 12
Completed | 12 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Overall: In Period 1, participants received a single oral dose of 18 milligram (mg) LY2216684, administered in either fasted or fed state. In Period 2, participants received a single oral dose of 18 mg LY2216684, administered in the alternative feeding state that was not used during Period 1 (fasted or fed). Periods were separated by a 7-day washout period.
Arm/Group | Overall
Number analyzed (Participants) | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.0 (12.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10
  Not Hispanic or Latino | 14
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 9
  White | 12
  More than one race | 3
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 24

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics: Area Under the Plasma Concentration-Time Curve From Time 0 to Infinity (AUC0-∞) of LY2216684
Description: The AUC for LY2216684 was calculated for LY2216684 administered in fed state (test) and LY2216684 administered in fasted state (reference). Geometric Least Squares (LS) means were calculated according to the following model: Log(PK) = sequence + period + treatment + subject + random error for AUC.
Time Frame: 0, 0.5, 1, 2, 3, 4, 5, 6, 8, 12, 24, 24, 48, 72 hours post dose
Population: All participants with a baseline observation and at least 1 post-baseline observation.
Measure: Least Squares Mean (90% Confidence Interval); unit: nanogram*hour/milliliter (ng*h/mL)
Groups:
- LY2216684 Administered in Fed State: Participants received a single oral dose of 18 mg LY2216684 in fed state.
- LY2216684 Administered in Fasted State: Participants received a single oral dose of 18 mg LY2216684 in fasted state.
Arm/Group | LY2216684 Administered in Fed State | LY2216684 Administered in Fasted State
Number analyzed (Participants) | 24 | 24
nanogram*hour/milliliter (ng*h/mL) | 871 [779 to 973] | 861 [771 to 962]
Statistical Analysis 1: Comparison: LY2216684 Administered in Fed State vs LY2216684 Administered in Fasted State; Test type: Superiority or Other; Mixed Models Analysis; Analyzed was a ratio of geometric LS means between the 2 treatment states (fed/fasted), and the 90% confidence interval for the ratio; Ratio of Geometric Least Squares Means = 1.01, 90% CI 2-sided [0.97 to 1.05]

2. Primary Outcome: Pharmacokinetics: Maximum Plasma Concentration (Cmax) of LY2216684
Description: The Cmax for LY2216684 was calculated for LY2216684 administered in fed state (test) and LY2216684 administered in fasted state (reference). Geometric LS means were calculated according to the following model: Log(PK) = sequence + period + treatment + subject + random error for Cmax.
Time Frame: 0, 0.5, 1, 2, 3, 4, 5, 6, 8, 12, 24, 24, 48, 72 hours post dose
Population: All participants with a baseline observation and at least 1 post-baseline observation.
Measure: Least Squares Mean (90% Confidence Interval); unit: nanogram/milliliter (ng/mL)
Arm/Group | LY2216684 Administered in Fed State | LY2216684 Administered in Fasted State
Number analyzed (Participants) | 24 | 24
nanogram/milliliter (ng/mL) | 66.04 [59.85 to 72.88] | 68.68 [62.24 to 75.78]
Statistical Analysis 1: Comparison: LY2216684 Administered in Fed State vs LY2216684 Administered in Fasted State; Test type: Superiority or Other; Mixed Models Analysis; Analyzed was a ratio of geometric LS means between the 2 treatments states (fed/fasted), and the 90% confidence interval for the ratio; Ratio of Geometric Least Squares Means = 0.96, 90% CI 2-sided [0.92 to 1.01]

3. Primary Outcome: Pharmacokinetics: Time to Maximum Plasma Concentration (Tmax) of LY2216684
Time Frame: 0, 0.5, 1, 2, 3, 4, 5, 6, 8, 12, 24, 24, 48, 72 hours post dose
Population: All participants with a baseline observation and at least 1 post-baseline observation.
Measure: Median (Full Range); unit: hours
Arm/Group | LY2216684 Administered in Fed State | LY2216684 Administered in Fasted State
Number analyzed (Participants) | 24 | 24
hours | 3.00 [1.00 to 6.00] | 2.00 [1.00 to 3.00]
Statistical Analysis 1: Comparison: LY2216684 Administered in Fed State vs LY2216684 Administered in Fasted State; Test type: Superiority or Other; p = 0.0031, Wilcoxon (Mann-Whitney); Analyzed were the median of paired differences between the 2 treatment states (fed versus fasted) and the 90% confidence interval; Median Difference (Final Values) = 1.00, 90% CI 2-sided [0.50 to 1.50]

ADVERSE EVENTS:
Arm/Group | LY2216684 Administered in Fed State | LY2216684 Administered in Fasted State
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/24
Other Adverse Events (participants affected / at risk) | 7/24 | 6/24
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LY2216684 Administered in Fed State (N=24) | LY2216684 Administered in Fasted State (N=24)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Asthenia (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 2 (2)
Scratch (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1)
Head discomfort (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 3 (3) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days